CLINICAL TRIAL: NCT06450119
Title: The Improvement of Cognition and Physical Function in Middle-aged and Older Adults With Cognitive Frailty: the Effectiveness of a Dual-task Training Program
Brief Title: The Effectiveness of a Dual-task Training Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huang, Hui-Chuan, Professor, School of Nursing, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N202304115
Record Dates: First submitted 2024-06-02; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Frailty; Cognitive Decline
Keywords: Cognitive frailty, Cognition, Dual-task training, Frailty
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- dual-task training (Experimental): walking and cognition training
  Interventions: Other: walking training; Other: cognition training
- walking training alone (Active Comparator): walking training
  Interventions: Other: walking training
- cognition training alone (Active Comparator): cognition training
  Interventions: Other: cognition training
- waiting list group (No Intervention): no intervention

INTERVENTIONS:
Other: walking training — The walking training alone group would receive walking training for 60 minutes twice weekly for twelve weeks.
  Arms: dual-task training; walking training alone
Other: cognition training — The cognition training alone group would receive cognition training for 60 minutes twice weekly for twelve weeks.
  Arms: cognition training alone; dual-task training

SUMMARY:
The purpose of this study is to explore the effect of a dual-task training intervention on cognitive function,physical function, depression symptoms and quality of life in middle-aged and elderly people with cognitive impairment. A Randomized experimental research design is conduced to recruited 196 middle-aged and elderly people: potentially reversible or reversible cognitive decline to attend this study. All participants are randomly allocated into dual-task training, walking training alone, and cognitive training alone and the waiting list control group. The measurements include: demographic and disease data, frailty symptoms (The FRAIL Scale ,Time up and go test ,Sit-to-stand test), cognitive function (Montreal Cognitive Assessment Scale Chinese version), depressive symptoms (Chinese version of Clinical Depression Symptom Assessment Scale) and life Quality (Taiwan's simplified version of the World Health Organization Quality of Life Questionnaire). The results of the study will use Generalized Liner Models and Pearson's product difference correlation analysis to confirm the impact of dual task training intervention on physical function, cognitive function, and depressive symptoms in middle-aged and elderly people with cognitive impairment effect on quality of life.

DETAILED DESCRIPTION:
A Randomized experimental research design is conduced to recruited 196 middle-aged and elderly people: potentially reversible or reversible cognitive decline to attend this study. All participants are randomly allocated into dual-task training, walking training alone, and cognitive training alone and the waiting list control group.

The dual task training group will receive 12 weeks of walking and cognitive training.

The walking training alone group will receive 12 wees of walking training. The cognitive training alone group will receive 12 weeks of cognitive training. Each session is 60 minutes and twice a week. The waiting list control group will not receive intervention activities. Outcomes are measured both before and after the intervention. The measurements include: demographic and disease data, frailty symptoms (The FRAIL Scale ,Time up and go test ,Sit-to-stand test), cognitive function (Montreal Cognitive Assessment Scale Chinese version), depressive symptoms (Chinese version of Clinical Depression Symptom Assessment Scale) and life Quality (Taiwan's simplified version of the World Health Organization Quality of Life Questionnaire). The results of the study will use Generalized Liner Models and Pearson's product difference correlation analysis to confirm the impact of the dual task training intervention on physical function, cognitive function, and depressive symptoms in middle-aged and elderly people with cognitive impairment effect on quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. age more than 50 years;
2. with physical frailty identified as The FRAIL Scale ≥1
3. subjective cognitive decline(subjective memory complain ≥3);
4. with literacy;
5. without regular exercise habits (<150 minutes/weekly);
6. without receiving cognitive training

Exclusion Criteria:

1. incapable of walking independent;
2. with diagnosis of cancer, dementia,neurological diseases (e.g., stroke, head injury, and brain tumor), psychiatric disorders (e.g.,depression, bipolar, and schizophrenia), cardiac infraction,and hemodialysis.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2024-06-03 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The FRAIL Scale | Baseline
  The FRAIL scale (short five-questions assessment of fatigue, resistance, aerobic capacity, illnesses and loss of weight) classified the patients into three categories: robust (score=0), pre-frailty (score=1-2), and frailty (score=3-5)
The FRAIL Scale | at 12 weeks after intervention
  The FRAIL scale (short five-questions assessment of fatigue, resistance, aerobic capacity, illnesses and loss of weight) classified the patients into three categories: robust (score=0), pre-frailty (score=1-2), and frailty (score=3-5)
Time up and go test | Baseline
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls
Time up and go test | at 12 weeks after intervention
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. scores of ten seconds or less indicate normal mobility, 11-20 seconds are within normal limits for frail elderly and disabled patients, and greater than 20 seconds means the person needs assistance outside and indicates further examination and intervention. A score of 30 seconds or more suggests that the person may be prone to falls
Sit-to-stand test | Baseline
  The score is the total number of stands within 30 second.
Sit-to-stand test | at 12 weeks after intervention
  The score is the total number of stands within 30 second.
cognitive function (Montreal Cognitive Assessment Scale Chinese version) | Baseline
  Montreal Cognitive Assessment Scale Chinese version is a 30-point test that assesses nine cognitive domains (executive function, language, orientation, calculation, conceptual thinking, memory, visual perception, naming and attention). MoCA for MCI detection were 19 in the low-level education group (≤6 years), 22 in the mid-level education group (7-12 years) and 24 in the high-level education group (>12 years), respectively.
cognitive function (Montreal Cognitive Assessment Scale Chinese version) | at 12 weeks after intervention
  Montreal Cognitive Assessment Scale Chinese version is a 30-point test that assesses nine cognitive domains (executive function, language, orientation, calculation, conceptual thinking, memory, visual perception, naming and attention). MoCA for MCI detection were 19 in the low-level education group (≤6 years), 22 in the mid-level education group (7-12 years) and 24 in the high-level education group (>12 years), respectively.

SECONDARY OUTCOMES:
depressive symptoms (Chinese version of Clinical Depression Symptom Assessment Scale) | Baseline
  The Chinese version of Clinical Depression Symptom Assessment Scale contains 18 items assessing all of the DSM-IV inclusion criteria for major depressive disorder as well as psychosocial impairment and quality of life.Total symptom scores on the scale range from 0 to 64. Empirically derived severity score ranges are 0-10 (nondepressed), 11-20 (minimal depression), 21-30 (mild depression), 31-45 (moderate depression), and 46-64 (severe depression).
depressive symptoms (Chinese version of Clinical Depression Symptom Assessment Scale) | at 12 weeks after intervention
  The Chinese version of Clinical Depression Symptom Assessment Scale contains 18 items assessing all of the DSM-IV inclusion criteria for major depressive disorder as well as psychosocial impairment and quality of life.Total symptom scores on the scale range from 0 to 64. Empirically derived severity score ranges are 0-10 (nondepressed), 11-20 (minimal depression), 21-30 (mild depression), 31-45 (moderate depression), and 46-64 (severe depression).
quality of life ( Taiwan's simplified version of the World Health Organization Quality of Life Questionnaire) | Baseline
  The Taiwan's simplified version of the World Health Organization Quality of Life Questionnaire is a 28-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (4 items), and environmental health (9 items). Higher scores indicates good quality of life.
quality of life ( Taiwan's simplified version of the World Health Organization Quality of Life Questionnaire) | at 12 weeks after intervention
  TheTaiwan's simplified version of the World Health Organization Quality of Life Questionnaire is a 28-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (4 items), and environmental health (9 items). Higher scores indicates good quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Huang, PhD, Principal Investigator — Taipei Medical University